CLINICAL TRIAL: NCT02638051
Title: Local Modulated Electro-Hyperthermia in Combination With Traditional Chinese Medicine Versus Intraperitoneal Chemoinfusion in Treatment of Peritoneal Carcinomatosis With Malignant Ascites: A Phase II Randomized Trial
Brief Title: Local mEHT + TCM Versus Intraperitoneal Chemoinfusion in Treatment of Malignant Ascites: Phase II RCT
Acronym: OTMA-RII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galenic Research Institute Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OT-CH-PCMA-14
Record Dates: First submitted 2015-12-17; First posted 2015-12-22 (Estimated); Results first posted 2016-03-28 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2015-12

CONDITIONS: Peritoneal Neoplasms; Ascites; Yang Deficiency; Yin Deficiency
Keywords: Peritoneal Carcinomatosis; Malignant Ascites; Modulated Electro-Hyperthermia; Traditional Chinese Medicine
MeSH Terms: conditions — Peritoneal Neoplasms; Ascites; Yang Deficiency; Yin Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Group (Experimental): Modulated Electro-Hyperthermia (mEHT): 150 Watt x 60 min/session every 2nd day for 4 weeks (14 sessions); TCM Herbal Decoction: Shi Pi Decoction administered orally twice a day (200 mL x 2) 30 min after breakfast and supper, for 4 weeks.
  Interventions: Device: Modulated Electro-Hyperthermia (mEHT); Dietary Supplement: TCM Herbal Decoction (Shi Pi)
- Control Group (Active Comparator): IPCI: CDDP (30-60 mg) with 5FU (500-600 mg/sqm of body surface), both dissolved in 100 mL of normal saline, after abdominal paracentesis and catheterization with following closed drainage of the ascites up to small amount of remaining liquid. After IPCI, the catheter occluded. Administered biweekly during four weeks of the course, totally two times.
  Interventions: Drug: IPCI (CDDP+5FU)

INTERVENTIONS:
Device: Modulated Electro-Hyperthermia (mEHT) — MEHT is a descendant of hyperthermia initially based on nano-thermal but not temperature-dependent effects of electromagnetic fields and special fractal modulation, whose effect could 3-4 times exceed the effect of the overall heating (macroscopic temperature elevation). MEHT does not require hyperthermia-range temperatures and could be performed safely without invasive thermal control. EHY-2000 local machine is used for mEHT in the trial.
  Other Names: Oncothermia
  Arms: Study Group
Dietary Supplement: TCM Herbal Decoction (Shi Pi) — Shi Pi Decoction can warm Yang, invigorate the spleen, promote Qi circulation to induce diuresis and treat Foot-Taiyin meridian in Gu Zhang.
  Other Names: Shi Pi Decoction
  Arms: Study Group
Drug: IPCI (CDDP+5FU) — Intraperitoneal chemoinfusion of CDDP (30-60 mg) and 5-fluorouracil (500-600 mg/sqm).
  Arms: Control Group

SUMMARY:
This trial studies efficacy and safety of combination of modulated electro-hyperthermia (mEHT) with Traditional Chinese Medicine (TCM) in treatment of peritoneal carcinomatosis with malignant ascites versus standard chemoinfusion (CDDP+5FU).

DETAILED DESCRIPTION:
Conservative treatment of peritoneal carcinomatosis with malignant ascites (PCMA) is based on chemoinfusion with its inherent toxicity. There is a strong demand for a safe and non-toxic method of treatment of PCMA. The new technology of modulated electro-hyperthermia (mEHT) has proven efficacy in many advanced cancers with minimal side effects and synergy with Traditional Chinese Medicine (TCM). TCM has a long history of application at advanced cancer as a symptomatic treatment and enhancer of the general resistance of the organism. Shi Pi Decoction is supposed to be the optimum co-treatment of PCMA according to principles of TCM. Intraperitoneal chemoinfusion (IPCI) with cisplatin and fluorouracil is a widespread standard treatment of PCMA in China. This randomized II phase trial studies efficacy and safety of combination of mEHT with TCM in treatment of PCMA versus standard IPCI (CDDP+5FU).

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed PC with malignant ascites.
* Karnofsky Performance Status (KPS) score ≥60%.
* Normal function of bone marrow.
* Predicted survival time >1 month.
* Written informed consent.

Exclusion Criteria:

* Surgery within 3 weeks or not full recovery of postoperative suture.
* Active bleeding or vascular occlusion in the mEHT treatment area.
* Emotional instability.
* Impossibility to place the patient into the mEHT machine.
* Metallic implants or replacements in the treatment area.
* Electronic implanted devices anywhere.
* Missing or damaged heat-sense nerves or other field-sensitive issues in the treatment area.
* Very low white blood cell count (<1.5×10(9)/L), agranulocytosis (<0.5×10(9)/L) or severe anemia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clifford LK Pang, PhD, Principal Investigator — Clifford Hospital
Locations (1):
- Clifford Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sangisetty SL, Miner TJ. Malignant ascites: A review of prognostic factors, pathophysiology and therapeutic measures. World J Gastrointest Surg. 2012 Apr 27;4(4):87-95. doi: 10.4240/wjgs.v4.i4.87. PMID 22590662
- [Background] Andocs G, Renner H, Balogh L, Fonyad L, Jakab C, Szasz A. Strong synergy of heat and modulated electromagnetic field in tumor cell killing. Strahlenther Onkol. 2009 Feb;185(2):120-6. doi: 10.1007/s00066-009-1903-1. Epub 2009 Feb 25. PMID 19240999
- [Background] Meggyeshazi N, Andocs G, Balogh L, Balla P, Kiszner G, Teleki I, Jeney A, Krenacs T. DNA fragmentation and caspase-independent programmed cell death by modulated electrohyperthermia. Strahlenther Onkol. 2014 Sep;190(9):815-22. doi: 10.1007/s00066-014-0617-1. Epub 2014 Feb 22. PMID 24562547
- [Background] Ling Y. Traditional Chinese medicine in the treatment of symptoms in patients with advanced cancer. Ann Palliat Med. 2013 Jul;2(3):141-52. doi: 10.3978/j.issn.2224-5820.2013.04.05. PMID 25842096
- [Background] Andocs G, Meggyeshazi N, Balogh L, Spisak S, Maros ME, Balla P, Kiszner G, Teleki I, Kovago C, Krenacs T. Upregulation of heat shock proteins and the promotion of damage-associated molecular pattern signals in a colorectal cancer model by modulated electrohyperthermia. Cell Stress Chaperones. 2015 Jan;20(1):37-46. doi: 10.1007/s12192-014-0523-6. Epub 2014 Jun 29. PMID 24973890
- [Background] Tsang YW, Huang CC, Yang KL, Chi MS, Chiang HC, Wang YS, Andocs G, Szasz A, Li WT, Chi KH. Improving immunological tumor microenvironment using electro-hyperthermia followed by dendritic cell immunotherapy. BMC Cancer. 2015 Oct 15;15:708. doi: 10.1186/s12885-015-1690-2. PMID 26472466
- [Background] Matharu G, Tucker O, Alderson D. Systematic review of intraperitoneal chemotherapy for gastric cancer. Br J Surg. 2011 Sep;98(9):1225-35. doi: 10.1002/bjs.7586. Epub 2011 Jun 6. PMID 21644239
- [Result] Pang CLK, Zhang X, Wang Z, Ou J, Lu Y, Chen P, Zhao C, Wang X, Zhang H, Roussakow SV. Local modulated electro-hyperthermia in combination with traditional Chinese medicine vs. intraperitoneal chemoinfusion for the treatment of peritoneal carcinomatosis with malignant ascites: A phase II randomized trial. Mol Clin Oncol. 2017 May;6(5):723-732. doi: 10.3892/mco.2017.1221. Epub 2017 Apr 10. PMID 28529748
- Available data/document: Clinical Study Report: 10.3892/mco.2017.1221 — https://www.spandidos-publications.com/mco/6/5/723?articleTypes=ARTICLE&articleTypes=REVIEW&fileTypes=LETTER_TO_THE_EDITOR&fileTypes=MANUSCRIPT&fileTypes=TABLE&fileTypes=IMAGE&fileTypes=LANG_EDIT — Pang CLK, Zhang X, Wang Z, Ou J, Lu Y, Chen P, Zhao C, Wang X, Zhang H, Roussakow SV. Local modulated electro-hyperthermia in combination with traditional Chinese medicine vs. intraperitoneal chemoinfusion for the treatment of peritoneal carcinomatosis with malignant ascites: A phase II randomized trial. Mol Clin Oncol. 2017;6:723-32,

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From January 3, 2014 to December 20, 2014, 260 patients were recruited in Clifford Hospital. They were randomly allocated in two groups with 130 patients in each group.
Pre-assignment Details: There was no any pre-assignment dropout or exclusion.
Groups:
- Control Group: IPCI: CDDP (30-60 mg) with 5FU (500-600 mg/sqm of body surface), both dissolved in 100 mL of normal saline, after abdominal paracentesis and catheterization with following closed drainage of the ascites up to small amount of remaining liquid. After IPCI, the catheter was occluded. Administered biweekly during four weeks of the course, totally two times.
  IPCI (CDDP+5FU): Intraperitoneal chemoinfusion of CDDP (30-60 mg) and 5-fluorouracil (500-600 mg/sqm).
Period: Overall Study
Arm/Group | Study Group | Control Group
Started | 130 | 130
Completed | 130 | 130
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group | Control Group | Total
Number analyzed (Participants) | 130 | 130 | 260
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.88 (12.43) | 56.07 (15.38) | 57.48 (14.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 61 | 133
  Male | 58 | 69 | 127
Region of Enrollment [Number; unit: participants]
  China | 130 | 130 | 260
Primary Disease [Number; unit: participants]
  Gastric Cancer | 22 | 24 | 46
  Colon Cancer | 34 | 37 | 71
  Rectal Cancer | 18 | 15 | 33
  Pancreatic Cancer | 13 | 8 | 21
  Endometrial Cancer | 9 | 5 | 14
  Ovarian Cancer | 11 | 16 | 27
  Liver Cancer | 23 | 25 | 48
Metastases [Number; unit: participants]
  Lungs | 23 | 20 | 43
  Liver | 32 | 35 | 67
  Celiac lymph nodes | 53 | 50 | 103
  Bones | 22 | 25 | 47
Stage [Number; unit: participants] — Peritoneal carcinomatosis itself is considered III stage; evidence of distant metastases means IV stage.
  participants
    I | 0 | 0 | 0
    II | 0 | 0 | 0
    III | 66 | 76 | 142
    IV | 64 | 54 | 118
Karnofsky Performance Score [Number; unit: participants] — KPS 90% - symptomatic patients with normal daily activity. KPS 80% - normal daily activity with effort. KPS 70% - limited daily activity (unable to work), complete self-care. KPS 60% - limited daily activity (unable to work), limited self-care (needs assistance), active >50% of daytime.
  KPS <60% (Perforce inactive (sits or lies) ≥50% of daytime) excluded.
  participants
    60 | 26 | 21 | 47
    70 | 50 | 47 | 97
    80 | 42 | 48 | 90
    90 | 12 | 14 | 26
CDDP (Intraperitoneal Chemoinfusion) Dose Per Session [Mean (Standard Deviation); unit: mg] | 0 (0) | 49.63 (10.19) | NA (NA) — CDDP applied in Control Group only, total result is not applicable
5-FU (Intraperitoneal Chemoinfusion) Dose Per Session [Mean (Standard Deviation); unit: mg/sqm] | 0 (0) | 548.5 (39.68) | NA (NA) — 5FU applied in Control Group only, total result is not applicable
Interventions [Median (Full Range); unit: sessions]
  mEHT | 14 [14 to 14] | 0 [0 to 0] | NA [NA to NA] — mEHT applied in Study Group only, total result is not applicable
  TCM | 28 [28 to 28] | 0 [0 to 0] | NA [NA to NA] — TCM applied in Study Group only, total result is not applicable
  IPCI | 0 [0 to 0] | 2 [2 to 2] | NA [NA to NA] — IPCI applied in Control Group only, total result is not applicable

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate (ORR) = Complete Remission (CR) + Partial Remission (PR)
  WHO criteria of therapeutic effect evaluation at malignant ascites:
  * Complete Remission (CR): complete absorption of ascites with no obvious regeneration for more than 1 month.
  * Partial Remission (PR): more than 50% reduction of ascites, with obvious relief of abdominal distention, with maintenance of less than moderate volume of ascites under ultrasound detection for more than 1 month.
  * No Change (NC): less than 50% reduction of ascites, or no obvious reduction of ascites under ultrasound detection, or even increase of ascites, with obvious abdominal distention.
Time Frame: 8 weeks after start of treatment (4 weeks on completion of treatment)
Measure: Number; unit: percentage of participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 130 | 130
percentage of participants | 77.7 | 63.8
Statistical Analysis 1: Comparison: Study Group vs Control Group; Applies to "Objective Response Rate (ORR)"; Test type: Superiority or Other; p = 0.0140, Chi-squared

2. Secondary Outcome: Adverse Events Rate (AER)
Description: Common Terminology Criteria for Adverse Events (CTCAE) (v4.03: June 14, 2010) U.S.DEPARTMENT OF HEALTH AND HUMAN SERVICES, National Institutes of Health, National Cancer Institute.
Time Frame: During 4 weeks of treatment course and 4 weeks after treatment
Measure: Number; unit: participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 130 | 130
participants
  All | 3 | 16
  Abdominal pain (Gr. I) | 3 | 5
  Gastrointestinal Reactions (Gr. I) | 0 | 3
  Damage of hepatic or renal function (Gr. I) | 0 | 2
  Bone marrow depression (Gr. I) | 0 | 6
Statistical Analysis 1: Comparison: Study Group vs Control Group; Applies to "All" Adverse Events rate; Test type: Superiority or Other; p = 0.0016, Chi-squared
Statistical Analysis 2: Comparison: Study Group vs Control Group; Applies to "Abdominal pain" rate; Test type: Superiority or Other; p > 0.05, Chi-squared
Statistical Analysis 3: Comparison: Study Group vs Control Group; Applies to "Gastrointestinal reactions"; Test type: Superiority or Other; p > 0.05, Chi-squared
Statistical Analysis 4: Comparison: Study Group vs Control Group; Applies to "Damage of hepatic or renal function"; Test type: Superiority or Other; p > 0.05, Chi-squared
Statistical Analysis 5: Comparison: Study Group vs Control Group; Applies to "Bone marrow depression"; Test type: Superiority or Other; p = 0.0215, Chi-squared

3. Secondary Outcome: Quality of Life (QoL)
Description: Karnofsky Performance Score Improvement Rate (KPS IR)
  * Improvement: increase of KPS for ≥10% after treatment.
  * Worsening: reduction of KPS for ≥10% after treatment.
  * NC: change of KPS for <10%.
Time Frame: 8 weeks after start of treatment (4 weeks on completion of treatment)
Measure: Number; unit: percentage of participants
Arm/Group | Study Group | Control Group
Number analyzed (Participants) | 130 | 130
percentage of participants
  Better QoL (KPS IR) | 49.2 | 32.3
  No Change | 40.8 | 52.3
  Worse QoL | 10 | 15.4
Statistical Analysis 1: Comparison: Study Group vs Control Group; Applies to "Better QoL"; Test type: Superiority or Other; p = 0.0053, Chi-squared
Statistical Analysis 2: Comparison: Study Group vs Control Group; Applies to "No Change"; Test type: Superiority or Other; p = 0.0527, Chi-squared
Statistical Analysis 3: Comparison: Study Group vs Control Group; Applies to "Worse QoL"; Test type: Superiority or Other; p > 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: 2 months
Description: The adverse events were accounted based on the objective data and voluntary testimonies of patients or through non-leading questions, and were timely recorded into the "Table of Adverse Events".
Arm/Group | Study Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/130 | 0/130
Other Adverse Events (participants affected / at risk) | 3/130 | 16/130
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Group (N=130) | Control Group (N=130)
Bone marow depression (Blood and lymphatic system disorders) | 0 (0) | 6 (6)
Abdominal Pain (Gastrointestinal disorders) | 3 (3) | 5 (5)
Gastrointestinal Reactions (Gastrointestinal disorders) | 0 (0) | 3 (3)
Damage of hepatic function (Hepatobiliary disorders) | 0 (0) | 1 (1)
Damage of renal function (Renal and urinary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
* Absence of the detailed peritoneal carcinomatosis characteristics.
* Absence of a survival analysis. These limitations are related to the restricted funding of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No